CLINICAL TRIAL: NCT00887354
Title: Comparison of the Effects of Teriparatide With Those of Risedronate on Lumbar Spine BMD (Bone Mineral Density) in Men and Postmenopausal Women With Low Bone Mass and a Recent Pertrochanteric Hip Fracture
Brief Title: A Study That Will Compare the Effect of Two Drugs on Participants With Low Bone Mass and a Recent Hip Fracture
Acronym: MOVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12400; B3D-EW-GHDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Osteoporosis
Keywords: Low bone mass; Recent pertrochanteric hip fracture
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Risedronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): 20 micrograms (mcg) a day by subcutaneous injection throughout study.
  Placebo oral tablets once a week, to match the active comparator weekly dose, during the double-blind, double-dummy phase only.
  Interventions: Drug: Teriparatide; Drug: Placebo; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Risedronate (Active Comparator): 35 milligrams (mg) risedronate sodium orally once weekly throughout study.
  Daily placebo injection, to match the daily experimental drug dose, during the double-blind, double-dummy phase only.
  Interventions: Drug: Risedronate; Drug: Placebo; Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Teriparatide — Administered subcutaneously
  Other Names: Forteo; LY333334
  Arms: Teriparatide
Drug: Risedronate — Administered orally
  Arms: Risedronate
Drug: Placebo — Weekly: Administered orally
  Daily: Administered subcutaneously
Dietary Supplement: Calcium — Approximately 500 to 1000 mg/day administered orally throughout study.
Dietary Supplement: Vitamin D — Approximately 800 International Units per day (IU/day) administered orally throughout study.

SUMMARY:
This study will evaluate whether teriparatide is superior to the active comparator in the change from baseline of lumbar spine BMD (bone mineral density) in men and postmenopausal women with low bone mass and a recent pertrochanteric hip fracture.

DETAILED DESCRIPTION:
The study has 3 periods: a screening phase, a double-blind, double-dummy treatment phase from the time of randomization to the 26 weeks visit, and an open-label treatment phase of approximately 12 month duration, where participants will continue treatment with the same study drug that they were randomized to.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women aged ≥50 who have sustained a unilateral, fracture of the trochanteric region
* Lumbar spine BMD and/or femoral neck BMD and/or total hip BMD measurement of the contra lateral hip at least 2.0 SDs (standard deviation) below the average bone mass for young women and men

Exclusion Criteria:

* Clinically significant abnormal laboratory values
* History of unresolved skeletal diseases that affect bone metabolism
* Polytrauma participants and participants with fractures at more than one site

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2009-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM eastern time (UTC/GMT-5hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb, Croatia
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Klatovy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viborg
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orléans
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Etienne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villeurbanne
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki, Greece
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexicali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oslo, Norway
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marbella
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set (FAS) is defined as all randomized participants receiving at least one dose of study drug with at least one post-baseline efficacy measure.
Groups:
- Teriparatide: 20 microgram (mcg) a day by subcutaneous (SC) injection throughout study.
  Calcium: Approximately 500 to 1000 milligram per day (mg/day) administered orally throughout study.
  Vitamin D: Approximately 800 International Units per day (IU/day) administered orally throughout study.
- Risedronate: 35 mg risedronate sodium orally once weekly throughout study.
  Calcium: Approximately 500 to 1000 mg/day administered orally throughout study.
  Vitamin D: Approximately 800 International Units per day (IU/day) administered orally throughout study.
Period: Treatment Phase (Week 0 to Week 26)
Arm/Group | Teriparatide | Risedronate
Started | 111 | 113
Received at Least 1 Dose of Study Drug | 106 | 110
Included in Full Analysis Set | 86 | 85
Completed | 60 | 65
Not Completed | 51 | 48
Not completed — Death | 0 | 1
Not completed — Sponsor Decision | 1 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 14 | 8
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Entry Criteria Not Met | 3 | 3
Not completed — Caregiver Decision | 1 | 2
Not completed — No efficacy data | 20 | 25
Not completed — Not Treated | 5 | 3
Period: Open Label Phase (Week 26 to Week 78)
Arm/Group | Teriparatide | Risedronate
Started | 60 | 65
Completed | 57 | 59
Not Completed | 3 | 6
Not completed — Death | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least one dose of study drug and with at least one post-baseline efficacy measure.
Groups:
- Teriparatide: 20 mcg a day by SC injection throughout study.
  Calcium: Approximately 500 to 1000 mg/day administered orally throughout study.
  Vitamin D: Approximately 800 International Units per day (IU/day) administered orally throughout study.
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Risedronate | Total
Number analyzed (Participants) | 86 | 85 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.2 (7.96) | 76.4 (7.47) | 76.8 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 66 | 132
  Male | 20 | 19 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 86 | 85 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 3 | 4 | 7
  Canada | 0 | 2 | 2
  Czech Republic | 8 | 12 | 20
  United States | 1 | 4 | 5
  Norway | 5 | 2 | 7
  Denmark | 13 | 9 | 22
  Italy | 16 | 10 | 26
  Mexico | 6 | 12 | 18
  France | 5 | 8 | 13
  Germany | 2 | 1 | 3
  Spain | 21 | 19 | 40
  United Kingdom | 1 | 0 | 1
  Austria | 1 | 0 | 1
  Ireland | 1 | 0 | 1
  Sweden | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine Areal Bone Mineral Density (BMD)
Description: Least squares (LS) means obtained from mixed model repeated measures analysis including as fixed effects treatment and time with interaction, further adjusted for baseline lumbar spine BMD, type of hip fracture (31-A1/31-A2) and glucocorticoids used at baseline (Yes/No).
Time Frame: Baseline, Week 78
Population: All randomized participants receiving at least one dose of study drug and with at least one post-baseline efficacy measure.
Measure: Least Squares Mean (Standard Error); unit: gram per square centimeter (g/cm^2)
Groups:
- Teriparatide: 20 mg per day by SC injection throughout study.
  Calcium: Approximately 500 to 1000 mg/day administered orally throughout study.
  Vitamin D: Approximately 800 International Units per day (IU/day) administered orally throughout study.
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 61 | 66
gram per square centimeter (g/cm^2) | 0.094 (0.0075) | 0.055 (0.0081)
Statistical Analysis 1: Comparison: Teriparatide vs Risedronate; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; LS Mean = 0.040, 95% CI 2-sided [0.025 to 0.055]

2. Secondary Outcome: Change in Lumbar Spine Areal Bone Mineral Density
Description: as for outcome 1
Time Frame: Baseline, Week 26; Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 61 | 66
g/cm^2
  Week 26 | 0.053 (0.0074) | 0.032 (0.0081)
  Week 52 | 0.078 (0.0074) | 0.044 (0.0081)

3. Secondary Outcome: Change in Areal Bone Mineral Density Measured at the Femoral Neck and Total Hip of the Non-Fractured Limb
Description: Femoral neck BMD: Least squares (LS) means obtained from mixed model repeated measures analysis including as fixed effects treatment and time with interaction, further adjusted for baseline femoral neck BMD and type of hip fracture (31-A1/31-A2) .
  Total hip BMD: Least squares (LS) means obtained from mixed model repeated measures analysis including as fixed effects treatment and time with interaction, further adjusted for baseline total hip BMD, type of hip fracture (31-A1/31-A2) and duration of prior bisphosphonate use.
Time Frame: Baseline, Week 26; Baseline, Week 52; Baseline, Week 78
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/cm^2
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 60 | 61
g/cm^2
  Total Hip 26 Weeks | -0.001 (0.0042) | -0.001 (0.0042)
  Total Hip 52 Weeks | 0.001 (0.0042) | -0.001 (0.0042)
  Total Hip 78 Weeks | 0.007 (0.0042) | 0.005 (0.0043)
  Femoral Neck 26 Weeks | 0.002 (0.0044) | -0.009 (0.0043)
  Femoral Neck 52 Weeks | -0.000 (0.0044) | -0.006 (0.0044)
  Femoral Neck 78 Weeks | 0.012 (0.0044) | -0.007 (0.0045)

4. Secondary Outcome: Change From Baseline in Physical Component Summary of the Short Form-36 (SF-36) Questionnaire
Description: SF-36 is a self-reported questionnaire consisting of 36 questions covering 8 health domains. Each domain was scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning. The physical component summary (PCS) has been constructed based on the 8 SF-36 domains and consist of the physical functioning, bodily pain, role-physical, and general health scales (range = 0 to 100, with higher scores indicating better health status for functioning). Least squares (LS) means obtained from mixed model repeated measures analysis including as fixed effects treatment and time with interaction, further adjusted for type of hip fracture (31-A1/31-A2) and adequate reduction (Yes/No).
Time Frame: Baseline, Week 6; Baseline, Week 12; Baseline, Week 18; Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 67 | 65
units on a scale
  Week 6 | 7.37 (1.065) | 5.10 (1.087)
  Week 12 | 11.32 (1.207) | 11.09 (1.208)
  Week 18 | 14.37 (1.256) | 12.81 (1.260)
  Week 26 | 16.34 (1.278) | 14.36 (1.258)

5. Secondary Outcome: Percentage of Participants Reporting Hip Pain in Modification of the Charnley's Pain Scale
Description: Self-reported hip pain scale in which 0=no pain; 1=pain is slight or intermittent, pain on starting to walk but getting less with normal activity; 2=pain occurs only after some activity, disappears quickly with rest; 3=pain is tolerable, permitting limited activity; 4=pain is severe on attempting to walk, prevents all activity; 5=pain is severe and spontaneous.
Time Frame: Baseline
Population: All randomized participants receiving at least one dose of study drug and having baseline Charnley's Pain Scale data.
Measure: Number; unit: percentage of participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 85 | 85
percentage of participants
  0-No pain | 9.4 | 8.2
  1- Pain slight or intermittent | 4.7 | 12.9
  2- Pain occurs only after some activity | 23.5 | 20.0
  3- Pain is tolerable | 36.5 | 38.8
  4- Pain severe on attempting to walk | 20.0 | 15.3
  5- Pain severe and spontaneous | 5.9 | 4.7

6. Secondary Outcome: Visual Analog Scale (VAS)
Description: Visual analog pain scale is a measurement instrument to measure the level of hip pain. Scores range from 0 to 100 millimeter (mm) with higher score indicating greater pain. Least squares (LS) means obtained from mixed model repeated measures analysis including as fixed effects treatment and time with interaction, further adjusted for type of fracture (31-A1/31-A2), type of reduction (open/close), use of opioids (Yes/No), use of non-steroidal anti-inflammatory drugs, adequate reduction (Yes/No) and interaction between treatment and adequate reduction.
Time Frame: 6, 12, 18, and 26 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 63 | 62
millimeter (mm)
  Week 6 | 16.44 (3.977) | 23.54 (4.443)
  Week 12 | 9.28 (4.048) | 19.24 (4.452)
  Week 18 | 6.90 (4.147) | 18.19 (4.508)
  Week 26 | 4.48 (4.128) | 13.74 (4.505)

7. Secondary Outcome: Timed "Up and Go" Test
Description: Timed "Up and Go" test measures, in seconds, the time taken by an individual to stand up from a standard chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down. Least squares (LS) means obtained from mixed model repeated measures analysis including as fixed effects treatment and time with interaction, further adjusted for age, type of fracture (31-A1/31-A2), type of reduction (open/close), type of walking aid, baseline SF-36 PCS and baseline Charnley's pain score.
Time Frame: 6, 12, 18, and 26 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds (sec)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 79 | 78
seconds (sec)
  Week 6 | 26.45 (1.090) | 32.38 (1.085)
  Week 12 | 20.13 (1.092) | 24.48 (1.086)
  Week 18 | 17.75 (1.093) | 21.14 (1.087)
  Week 26 | 16.69 (1.095) | 19.91 (1.088)

ADVERSE EVENTS:
Description: Received at least one dose of study drug.
Arm/Group | Teriparatide | Risedronate
Serious Adverse Events (participants affected / at risk) | 21/106 | 27/110
Other Adverse Events (participants affected / at risk) | 53/106 | 47/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=106) | Risedronate (N=110)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Device breakage (General disorders) | 0 (0) | 1 (1)
Device failure (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 9 (9)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Teriparatide (N=106) | Risedronate (N=110)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (6) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7) | 4 (7)
Viral infection (Infections and infestations) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (8) | 5 (5)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (3)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1/23 (1)
Vulval ulceration (Reproductive system and breast disorders) | 0 (0) | 1/87 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1/81 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less